CLINICAL TRIAL: NCT07383441
Title: Phase III Double Blinded Trial of Immune-Based Therapy With a Live Biotherapeutic MO-03 or Placebo for Frontline Therapy of Advanced Clear Cell Renal Cell Carcinoma [BioFront Trial]
Brief Title: Adding Biotherapy or Placebo to Standard Treatment for Advanced Kidney Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S2419; NCI-2026-00080 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S2419 (Other: SWOG); S2419 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Advanced Clear Cell Renal Cell Carcinoma; Metastatic Clear Cell Renal Cell Carcinoma; Stage III Renal Cell Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma; Carcinoma, Renal Cell | interventions — Axitinib; Specimen Handling; cabozantinib; Ipilimumab; CTLA-4 Antigen; lenvatinib; Magnetic Resonance Spectroscopy; Nivolumab; Hyaluronoglucosaminidase; pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Double blinded trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (MO-03, SOC immunotherapy) (Experimental): See Detailed Description
  Interventions: Drug: Axitinib; Procedure: Biospecimen Collection; Procedure: Bone Scan; Drug: Cabozantinib; Drug: Clostridium butyricum CBM 588 Probiotic Strain; Procedure: Computed Tomography; Biological: Ipilimumab; Drug: Lenvatinib; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Drug: Nivolumab and Recombinant Human Hyaluronidase; Biological: Pembrolizumab
- Arm 2 (placebo, SOC immunotherapy) (Placebo Comparator): See Detailed Description
  Interventions: Drug: Axitinib; Procedure: Biospecimen Collection; Procedure: Bone Scan; Drug: Cabozantinib; Procedure: Computed Tomography; Biological: Ipilimumab; Drug: Lenvatinib; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Drug: Nivolumab and Recombinant Human Hyaluronidase; Biological: Pembrolizumab; Drug: Placebo Administration

INTERVENTIONS:
Drug: Axitinib — Given PO
  Other Names: AG 013736; AG-013736; AG013736; Inlyta
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Drug: Cabozantinib — Given PO
Drug: Clostridium butyricum CBM 588 Probiotic Strain — Given PO
  Other Names: C. butyricum CBM 588 Probiotic Strain; C. butyricum MIYAIRI Strain; C. butyricum Strain MIYAIRI 588; CBM 588; CBM588; Clostridium butyricum MIYAIRI 588; Clostridium butyricum MIYAIRI 588 Probiotic Strain; CLOSTRIDIUM BUTYRICUM MIYAIRI 588 STRAIN; MIYAIRI 588; MIYAIRI 588 Strain of C. butyricum
  Arms: Arm 1 (MO-03, SOC immunotherapy)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
Drug: Lenvatinib — Given PO
  Other Names: E 7080; E-7080; E7080; ER-203492-00; Multi-Kinase Inhibitor E7080
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
Drug: Nivolumab and Recombinant Human Hyaluronidase — Given SC
  Other Names: Hyaluronidase-nvhy and Nivolumab; Hyaluronidase/Nivolumab; Nivolumab and Hyaluronidase-nvhy; Nivolumab and rHuPH20; Nivolumab/Recombinant Human Hyaluronidase; Nivolumab/rHuPH20; Opdivo Qvantig
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
Drug: Placebo Administration — Given PO
  Arms: Arm 2 (placebo, SOC immunotherapy)

SUMMARY:
This phase III trial compares the effect of adding live biotherapy, MO-03, to standard of care (SOC) immunotherapy, including ipilimumab, nivolumab, axitinib, pembrolizumab, cabozantinib, and lenvatinib, to SOC immunotherapy alone in treating patients with clear cell renal cell cancer that may have spread from where it first started (primary site) to nearby tissue, lymph nodes, or distant parts of the body (advanced) or that has spread from where it first started to other places in the body (metastatic). Studies have shown that gut health (the gut microbiome) may impact the effectiveness of immunotherapy. The microbiome includes all of the bacteria and organisms naturally found in the digestive tract. MO-03, a type of biotherapy, contains material from living organisms that may help keep the digestive tract healthy and may help to increase the effect of immunotherapy. Immunotherapy with monoclonal antibodies, such as ipilimumab, nivolumab, pembrolizumab, may help the body's immune system attack the tumor, and may interfere with the ability of tumor cells to grow and spread. Axitinib, cabozantinib, and lenvatinib are a type of angiogenesis inhibitor and tyrosine kinase inhibitor (TKI) that block certain proteins which may help keep tumor cells from growing and may also help prevent the growth of new blood vessels that tumors need to grow. Adding MO-03 to SOC immunotherapy may be more effective than SOC immunotherapy alone in treating patients with advanced or metastatic clear cell renal cell cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare investigator assessed progression-free survival of participants with advanced clear cell renal cell carcinoma (ccRCC) randomized to standard of care immunotherapy (IO)-based combination regimen plus placebo versus IO-based combination regimen plus clostridium butyricum CBM 588 probiotic strain (MO-03) in an intent-to-treat analysis.

SECONDARY OBJECTIVES:

I. For the safety run-in: To assess the safety of MO-03 when added to each of the following standard frontline treatment regimens for advanced renal cell carcinoma: cabozantinib/nivolumab, axitinib/pembrolizumab (MK-3475) and lenvatinib/pembrolizumab (MK-3475) in the first 50 randomized patients after receiving at least two cycles of treatment.

II. To compare investigator assessed Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 response (confirmed and unconfirmed complete response and partial response) between the study arms.

III. To compare overall survival (OS) between the study arms. IV. To compare investigator assessed progression free survival (PFS) rates between the study arms at 12 months and at 24 months.

V. To evaluate the qualitative and quantitative toxicities between the study arms.

ADDITIONAL OBJECTIVES:

I. To compare time to subsequent systemic therapy between the study arms. II. To evaluate the potential impact of concomitant medications, specifically antibiotics, proton pump inhibitors (PPI) and steroids, on the activity of MO-03 in combination with standard immune checkpoint inhibitors (ICI) based regimen.

TRANSLATIONAL MEDICINE BANKING OBJECTIVE:

I. To bank archival tissue, blood and stool samples for future contemporary translational studies.

OUTLINE: Patients are randomized to 1 of 2 arms and are assigned to 1 of 4 regimens based on risk status.

ARM 1: Patients receive MO-03 orally (PO) twice daily (BID) on days 1-42 of each cycle. Cycles repeat every 42 days for up to 3 years in the absence of disease progression or unacceptable toxicity. In addition, intermediate or poor-risk patients also receive SOC immunotherapy regimens 1, 2, 3, or 4 and favorable risk patients receive SOC immunotherapy regimens 2, 3, or 4.

ARM 2: Patients receive placebo PO BID on days 1-42 of each cycle. Cycles repeat every 42 days for up to 3 years in the absence of disease progression or unacceptable toxicity. In addition, intermediate or poor-risk patients also receive SOC immunotherapy regimens 1, 2, 3, or 4 and favorable risk patients receive SOC immunotherapy regimens 2, 3, or 4.

REGIMEN 1: Patients receive SOC ipilimumab intravenously (IV) over 30-90 minutes and nivolumab IV or nivolumab and recombinant human hyaluronidase subcutaneously (SC) every 21 days for up to 4 infusions in the absence of disease progression or unacceptable toxicity. After completing 4 infusions, patients continue to receive nivolumab IV or nivolumab and recombinant human hyaluronidase SC every 14 or 28 days in the absence of disease progression or unacceptable toxicity.

REGIMEN 2: Patients receive SOC axitinib PO BID for up to 3 years in the absence of disease progression or unacceptable toxicity. Patients also receive SOC pembrolizumab IV every 21 or 42 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

REGIMEN 3: Patients receive SOC cabozantinib PO once daily (QD) for up to 3 years in the absence of disease progression or unacceptable toxicity. Patients also receive SOC nivolumab IV or nivolumab and recombinant human hyaluronidase SC every 14 or 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

REGIMEN 4: Patients receive SOC lenvatinib PO QD for up to 3 years in the absence of disease progression or unacceptable toxicity. Patients also receive SOC pembrolizumab IV every 21 or 42 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

All patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI) and blood sample collection throughout the study. Additionally, patients with suspected bone metastasis may undergo bone scan throughout the study and patients with suspected brain metastasis may undergo brain MRI throughout the study

After completion of study treatment, patients are followed every 6 months for the first 2 years then once a year for years 3-5.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed renal cell carcinoma (RCC) with clear cell component that is advanced (not amenable to curative surgery or radiation therapy) or metastatic RCC at the time of registration on study
* Participants must have measurable/evaluable disease by RECIST 1.1 criteria. Participants with only bone metastases or only pleural effusions are considered evaluable disease and are eligible
* Participants with new or progressive brain metastases (active brain metastases) or leptomeningeal disease must not require immediate central nervous system (CNS) specific treatment at the time of study registration or anticipated treatment during the first cycle of therapy
* Participants must not be currently enrolled or plan to participate in treatment studies while enrolled on this study
* Participants must not plan to take any over the counter probiotic supplements at time of study registration and while on protocol treatment

  * NOTE: Vitamin and electrolyte or mineral supplements are permitted
* Participants must not have had prior systemic therapy for advanced or metastatic RCC or any treatment with immune based combination therapy

  * NOTE: Participants can have prior neo/adjuvant treatment with an anti-PD-1, anti-PD-L1, and/or anti-CTLA-4 antibody or other therapies for any current or prior malignancy if > 12 months prior to registration
* Participants must not be receiving steroid replacement therapy for adrenal insufficiency greater than 50 mg daily of hydrocortisone or prednisone equivalent dose at the time of registration
* Participants must not require the use of systemic corticosteroids > 10 mg/day of prednisone or its equivalent for any reason other than replacement therapy for adrenal insufficiency
* Participants must not have received any systemic antibiotics within 7 days prior to registration

  * NOTE: Uncontrolled infections must be completely resolved
* Participants must be ≥ 18 years old at the time of registration
* Participants must have a Zubrod performance status 0-2 within 28 days of registration
* Participants must be able to safely receive at least one of the standard of care regimens, per the current Food and Drug Administration (FDA)-approved package inserts, treating investigator's discretion, and institutional guidelines

  * NOTE: Participants with favorable risk as defined by the International Metastatic RCC Database Consortium (IMDC) must plan to receive one of the TKI+ immunotherapy treatment combinations. They are not able to receive regimen 1 (ipilimumab + nivolumab) for this study
* Participants must be able to swallow and retain oral medications and have no known gastrointestinal disorders likely to interfere with absorption of oral medications
* Participants must have serum creatinine ≤ 2 x ULN (upper limit of normal). This specimen must have been drawn and processed within 28 days prior to registration
* Hemoglobin ≥ 8 g/dL (within 28 days prior to registration)
* Leukocytes ≥ 3 x 10^3/uL (within 28 days prior to registration)
* Absolute neutrophil count ≥ 1.5 x 10^3/uL (within 28 days prior to registration)
* Platelets ≥ 100 x 10^3/uL (within 28 days prior to registration)
* Total bilirubin ≤ institutional upper limit of normal (ULN) unless history of Gilbert's disease (within 28 days prior to registration) Participants with history of Gilbert's disease must have total bilirubin ≤ 5 x institutional ULN
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 3 x institutional ULN (< 5 x institutional ULN if liver metastases are present) (within 28 days prior to registration)
* Participants must have alkaline phosphate measured as a part of the liver function assessment within 28 days prior to registration
* Participants must have albumin corrected calcium measured within 28 days prior to registration
* Participants with a history human immunodeficiency virus (HIV)-infection must be on effective anti-retroviral therapy at registration and have undetectable viral load on the most recent test results obtained within 6 months prior to registration
* Participants with a history of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load while on suppressive therapy on the most recent test results obtained within 6 months prior to registration
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. Participants currently being treated for HCV infection must have undetectable HCV viral load test on the most recent test results obtained within 6 months prior to registration
* Participants must not have uncontrolled blood pressure and hypertension within 28 days prior to registration
* Participants must not have a prior or concurrent malignancy whose natural history or treatment (in the opinion of the treating physician) has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Participants must not have any known history of an autoimmune disease that prohibits the use of immune checkpoint therapy
* Participants must not be pregnant or nursing (nursing includes breast milk fed to an infant by any means, including from the breast, milk expressed by hand, or pumped). Individuals who are of reproductive potential must have agreed to use an effective contraceptive method with details provided as a part of the consent process. A person who has had menses at any time in the preceding 12 consecutive months or who has semen likely to contain sperm is considered to be of "reproductive potential." In addition to routine contraceptive methods, "effective contraception" also includes refraining from sexual activity that might result in pregnancy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) including hysterectomy, bilateral oophorectomy, bilateral tubal ligation/occlusion, and vasectomy with testing showing no sperm in the semen
* Participants must be offered the opportunity to participate in specimen banking
* Participants who have the ability to complete questionnaires in English or Spanish must be offered the opportunity to participate in the patient-reported outcome study
* NOTE: As a part of the OPEN registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system.

  * Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines
  * For participants with impaired decision-making capabilities, legally authorized representatives may sign and give informed consent on behalf of study participants in accordance with applicable federal, local, and Central Institutional Review Board (CIRB) regulations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 718 (Estimated)
Dates: Start 2026-06-10 (Estimated); Primary Completion 2033-01-31 (Estimated); Study Completion 2034-01-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From date of randomization to date of first documentation of progression, or death due to any cause, assessed up to 5 years
  A Cox model will be used to test the treatment hazard ratio with stratification factors in the model as covariates for the futility and efficacy interim analyses and the final analysis.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) (Safety run-in) | During the first 12 weeks (2 cycles [cycle length =42 days])
  Will be assessed according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. The rate and severity of toxicities on the active arm will be compared to the placebo arm to provide context for the background rate of toxicities attributable to the standard of care regimens.
Overall survival | From date of randomization to date of death due to any cause, assessed up to 5 years
  Will report the hazard ratio and 95% confidence interval for blinded study agent with respect to overall survival with stratification in the Cox model for the stratification factors.
PFS rates between the study arms | At 12 and 24 months
  Estimates of treatment effect and the corresponding 95% confidence interval will be provided for the PFS endpoint for sex, race, and ethnicity.
Incidence of AEs between study arms | Up to 90 days after last dose of study treatment
  Will be assessed according to the NCI CTCAE v 5.0. The rate and severity of toxicities on the active arm will be compared to the placebo arm to provide context for the background rate of toxicities attributable to the standard of care regimens.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Barata, Principal Investigator — SWOG Cancer Research Network